CLINICAL TRIAL: NCT05557071
Title: Increasing Physical Activity Among Early Career Professionals: A Feasibility Trial of an Online Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Professor, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-0412
Record Dates: First submitted 2022-09-18; First posted 2022-09-27 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Health Promotion; Physical Activity
Keywords: Emotion Regulation; Intention-behaviour Gap; Early Career Professionals
MeSH Terms: conditions — Motor Activity; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): An online, asynchronous, self-paced, 6-week long, physical activity intervention.
  Interventions: Behavioral: Digital Health Behaviour Change Platform
- Control (No Intervention): A waitlist control; continue with life/activity as usual. Control participants will receive access to the intervention at 6 weeks following all measurements.

INTERVENTIONS:
Behavioral: Digital Health Behaviour Change Platform — Participants will gain access to 6 weekly lessons.
  A series of 6 weekly educational modules including information on psychosocial determinants of physical activity engagement, adherence and maintenance, as well as corresponding behaviour change techniques and a number of other tools and strategies, such as reflection activities, quizzes, and worksheets. Mini podcasts are available to supplement the concepts introduced in the modules. The content is tailored for early career professionals. There will be an emphasis on tactics (e.g., mindfulness, acceptance, emotion regulation) to assist with overcoming incidental affect.
  Arms: Intervention

SUMMARY:
Physical activity promotion remains a public health priority and accessible and scalable interventions are needed. Early career professionals are at-risk for inactivity and therefore a critical target for physical activity promotion. An online delivery format made up of web-based lessons and podcasts meets accessibility needs for this time-pressed population and has strong potential for reach.

This study explores the feasibility of a theory-based intervention which accounts for action control, namely by leveraging the the Multi-Process Action Control framework (M-PAC) and targeting factors such as incidental affect (e.g., work-related stress) through emotion regulation strategies grounded in the principles of Acceptance and Commitment Therapy.

The primary objective of this study is to examine the feasibility and acceptability of a 6-week web-based physical activity behaviour change program for early career professionals. Primary outcomes include rates of recruitment, attention, adherence as well as study satisfaction and intervention acceptability. Secondary measures will include physical activity and emotion regulation. Additional measures will explore Multi-Process Action Control constructs, perceived stress, applied mindfulness, action and acceptance, and valued living.

DETAILED DESCRIPTION:
BACKGROUND

Despite the well-established physical and psychological benefit of physical activity, much of the population is not meeting recommended guidelines. Critical life transitions have been linked to physical activity decline and it follows that targeting those in transition is prudent. Early career professionals are one such critical demographic. Given the stress, demands, and time constraints that come with shifting to the workforce, it can be difficult to follow through on physical activity intentions. As such, an intervention designed to incorporate intention translation, mitigate incidental affect, and foster emotion regulation is warranted. This study will examine the feasibility of an accessible online intervention. Qualitative analysis will assist with refining the intervention and the protocol. Progression criteria will be used to determine whether revisions should be considered before proceeding to a definitive randomized controlled trial.

TARGET POPULATION

Early career professionals, operationalized as adults aged 25-44 and working at a desk-based job.

DESIGN

An open parallel feasibility randomized controlled trial will compare an online intervention condition to a waitlist control condition. This study features a controlled baseline with a post-intervention (6 weeks) evaluative design with an embedded qualitative and quantitative process evaluation.

INTERVENTION

Participants will be randomized to 1) a waitlist control group and 2) and Online Platform Intervention group.

Condition one: Waitlist control group representing the comparator. The control group will complete the baseline and final questionnaires. Following study completion, this group has the option of gaining access to the online platform for their own benefit.

Condition two: Intervention group. Those in the intervention condition will gain access to the online platform after completing a baseline questionnaire. Participants will engage in a self-guided 6 week program made up of weekly lessons. A 'booster session' will be offered at 3 weeks to check in regarding progress and engagement. A follow-up survey will be completed at 6 weeks, post-intervention. Participants will be invited to complete a qualitative semi-structured exit interview following final questionnaire completion.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults, aged 25-44, living in Canada, currently employed at least part-time in a desk-based job, currently not meeting physical activity guidelines, no contraindications to safely increase physical activity, access to the internet and a device to support the e-health application
* Report no contraindications to physical activity (based on the completion of the Physical Activity Readiness Questionnaire administered at screening)

Exclusion Criteria:

* No internet access, unable to speak/read English, meeting physical activity guidelines, existing chronic medical condition making them at risk of injury or ill health from increased physical activity
* No exclusion criteria for sex, gender, medications, race or religion will be applied.

Ages: 25 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate (monthly) | 4 months (at study completion)
  Primary outcome related to trial feasibility
Participant retention | 6 weeks
  Primary outcome related to trial feasibility
Adherence and engagement | 6 Weeks
  Primary outcome related to trial feasibility
Study satisfaction and acceptabiity | 6 Weeks
  Primary outcome related to trial acceptability

SECONDARY OUTCOMES:
Self-reported physical activity | 6 weeks
  measured using the Godin Leisure-Time Exercise Questionnaire (GLTEQ)
Emotion regulation | 6 weeks
  Adapted from DERS-16 (Bjureberg et al., 2016)

OTHER OUTCOMES:
Multi-Process Action Control constructs | 6 weeks
  Exploratory outcomes and manipulation checks
ACT Constructs | 6 weeks
  Exploratory outcomes and manipulation checks
Applied Mindfulness | 6 weeks
  Exploratory outcomes and manipulation checks

CONTACTS AND LOCATIONS:
Overall Officials: Stina J Grant, BA, Study Director — University of Victoria; Ryan E Rhodes, PhD, Principal Investigator — University of Victoria
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No